CLINICAL TRIAL: NCT05950087
Title: Study on the Relationship Between Plasma MRD and cfDNA HPV and the Efficacy and Prognosis of Locally Advanced Cervical Cancer After Concurrent Chemoradiotherapy
Status: Recruiting | Type: Observational
Sponsor: Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: (2023)089
Record Dates: First submitted 2023-06-09; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Concurrent chemoradiotherapy — Concurrent chemoradiotherapy

SUMMARY:
Cervical cancer CC is the most common malignant tumor in the female reproductive system, seriously endangering women's health and life, and is one of the leading causes of death for women worldwide.Globally, HPV causes about 85% of cervical cancers and about 60% of oropharyngeal cancers, causing more than 500,000 cancers each year.ctDNA is a potential biomarker because it contains tumor-specific genetic and epigenetic abnormalities that can be used in cancer diagnosis and prognosis prediction.MRD is considered a promising prognostic marker that can be used to identify individuals at increased risk of recurrence and individuals who may benefit from treatment.The expression level of MRD and plasma HPV before and after radiotherapy and chemotherapy for cervical cancer was analyzed by liquid biopsy ctDNA detection technology, which predicted the efficacy of cervical cancer radiotherapy and chemotherapy, which was helpful for monitoring and estimating the risk of disease recurrence after cervical cancer radiotherapy and chemotherapy, and verified the expression of MRD and plasma HPV as the basis for adjuvant chemotherapy after cervical cancer radiotherapy and the basis for optimal chemotherapy time node selection.

DETAILED DESCRIPTION:
Current treatments for cervical cancer include surgery, radiotherapy, chemotherapy, and immunotherapy. However,5 year survival remains unsatisfactory because most patients with cervical cancer are typically diagnosed locally advanced or have distant lymph node metastases.HPV can integrate its own genome into the host genome by disrupting the open reading frame of the E2 gene and increase the expression of the E6 and E7 genes. The p53 protein of the host cell is degraded by the production of the E6 virulent protein, which inactivates the pRb protein that controls the cell cycle, thereby cancerizing the entire host cell [6]. According to TCGA 2017 data, HPV integration into the host genome was found in more than 80% of HPV-positive cervical cancer patients. Han K et al. found that HPV testing can assess the prognosis of cervical cancer patients.Circulating tumor DNA (ctDNA), circulating tumor cells (CTCs), circulating tumor RNA (ctRNA), exosomes, proteins, and metabolites that are liquid biopsy analytes can be identified using biomarkers such as somatic point mutations, deletions, amplification, gene fusion, DNA methylation markers, miRNAs, proteins, or metabolites.Minimal tumor residual (MRD) refers to the residual tumor cells or biomarkers in the body after local or systemic cancer treatment, the activation of which can promote tumor metastasis and recurrence, also known as minimal residual disease, measurable residual disease, and molecular residual disease.Recently, the use of ctDNA analysis to determine MRD in solid tumors after intention-to-treat treatment and before clinical or radiological disease recurrence has shown significant therapeutic promise. In addition, MRD identification by ctDNA analysis correlates with poor prognosis in patients with malignant tumors.This project will use liquid biopsy ctDNA detection technology to analyze the expression level of MRD and plasma HPV before and after radiotherapy and chemotherapy for cervical cancer, predict the efficacy of radiotherapy and chemotherapy for cervical cancer, help monitor and estimate the risk of disease recurrence after radiotherapy and chemotherapy for cervical cancer, verify the expression of MRD and plasma HPV as the basis for adjuvant chemotherapy after radiotherapy and chemotherapy for cervical cancer and the basis for the selection of the optimal chemotherapy time, so as to provide clinically useful tumor markers for cervical cancer patients and reduce the mortality rate of cervical cancer.

ELIGIBILITY:
Inclusion criteria

* Age: ≥ 18 years old, ≤ 75 years old.
* Pathological histologic confirmation of cervical cancer.
* Imaging or PET/CT examination can be performed to understand the tumor and complete all follow-up.
* Measurable lesions before treatment.
* Good physical condition: ECOG score 0-1 (or KPS score 70-100).
* Estimated survival≥ 6 months.
* The baseline blood routine and biochemical indexes before radiotherapy and chemotherapy met the following standards: hemoglobin ≥ 80g/L, absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet ≥ 100×109/L, ALT, AST ≤ 2.5 times the normal upper limit; Serum albumin ≥ 30 g/L.
* There are three preoperative items: if the patient has syphilis, plum repellent therapy is required before treatment.
* The patient has no history of allergy to rubber products.
* Cardiopulmonary function is basically normal

Exclusion Criteria:

* Those who are allergic to rubber products.
* Those with severe acute infection and uncontrolled or purulent and chronic infection wounds that do not heal, chronic hepatitis B active stage, active tuberculosis, syphilis outbreak and AIDS.
* Patients with pre-existing severe heart disease, including: congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and intractable hypertension.
* Those with neurological or psychiatric diseases or mental disorders that are not easy to control, poor compliance, unable to cooperate with and describe treatment responses, uncontrolled primary brain tumors or central nervous system metastases, and those with obvious cranial hypertension signs or neuropsychiatric symptoms.
* with malignant serous effusion.
* History of severe enteritis and cystitis, bleeding, intestinal perforation, rectovaginal fistula, rectoval bladder fistula, etc.
* Those who have participated in other clinical trials.
* Other situations in which the investigator believes that the subject is not suitable to participate in this experiment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed cervical cancer patients who initially visited Guizhou Provincial People's Hospital from November 2022 to November 2024
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression levels of MRD | Before chemoradiotherapy
  Blood collected by patients prior to concurrent chemoradiotherapy were tested to observe the expression levels of MRD
Positive expression of plasma HPV | Before chemoradiotherapy
  Tissue samplescollected by patients prior to concurrent chemoradiotherapy were tested to observe the positive expression of plasma HPV
Expression levels of MRD | During concurrent chemoradiotherapy, up to 6 weeks
  Blood collected in concurrent chemoradiotherapy were examined to observe the expression levels of MRD
Positive expression of plasma HPV | During concurrent chemoradiotherapy,up to 6 weeks
  Tissue samples collected in concurrent chemoradiotherapy were examined to observe the positive expression of plasma HPV
Expression levels of MRD | 4 weeks after the end of concurrent chemoradiotherapy
  Blood collected 4 weeks after the end of concurrent chemoradiotherapy were tested to observe the expression levels of MRD
Positive expression of plasma HPV | 4 weeks after the end of concurrent chemoradiotherapy
  Tissue samples collected 4 weeks after the end of concurrent chemoradiotherapy were tested to observe the positive expression of plasma HPV
Expression levels of MRD | 12 weeks after the end of concurrent chemoradiotherapy
  Blood collected 12 weeks after the end of concurrent chemoradiotherapy were tested to observe the expression levels of MRD
Positive expression of plasma HPV | 12 weeks after the end of concurrent chemoradiotherapy
  Blood and tissue samples collected 12 weeks after the end of concurrent chemoradiotherapy were tested to observe the positive expression of plasma HPV
Expression levels of MRD | 24 weeks after the end of concurrent chemoradiotherapy
  Blood and tissue samples collected by patients 24 weeks after the end of concurrent chemoradiotherapy were tested to observe the expression levels of MRD
Positive expression of plasma HPV | 24 weeks after the end of concurrent chemoradiotherapy
  Blood and tissue samples collected by patients 24 weeks after the end of concurrent chemoradiotherapy were tested to observe the positive expression of plasma HPV

CONTACTS AND LOCATIONS:
Locations (1):
- Yong Li, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT05950087/Prot_000.pdf